CLINICAL TRIAL: NCT05356195
Title: A Phase 3 Study to Evaluate the Safety and Efficacy of a Single Dose of CTX001 in Pediatric Subjects With Transfusion-Dependent β-Thalassemia
Brief Title: Evaluation of Safety and Efficacy of CTX001 in Pediatric Participants With Transfusion-Dependent β-Thalassemia (TDT)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: CRISPR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX21-CTX001-141; 2021-002172-39 (EudraCT Number)
Record Dates: First submitted 2022-04-07; First posted 2022-05-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-02

CONDITIONS: Beta-Thalassemia; Thalassemia; Genetic Diseases, Inborn; Hematologic Diseases; Hemoglobinopathies
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Genetic Diseases, Inborn; Hematologic Diseases; Hemoglobinopathies | interventions — exagamglogene autotemcel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX001 (Experimental): CTX001 (autologous CD34+ hHSPCs modified with CRISPR-Cas9 at the erythroid lineage-specific enhancer of the BCL11A gene). Participants will receive single infusion of CTX001 through central venous catheter.
  Interventions: Biological: CTX001

INTERVENTIONS:
Biological: CTX001 — Administered by intravenous infusion following myeloablative conditioning with busulfan.
  Other Names: Exagamglogene autotemcel; Exa-cel

SUMMARY:
This is a single-dose, open-label study in pediatric participants with TDT. The study will evaluate the safety and efficacy of autologous CRISPR-Cas9 modified CD34+ human hematopoietic stem and progenitor cells (hHSPCs) (CTX001).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of TDT as defined by:

  * Documented homozygous or compound heterozygous β-thalassemia including β-thalassemia/hemoglobin E (HbE). Participants can be enrolled based on historical data, but a confirmation of the genotype using the study central laboratory will be required before busulfan conditioning
  * History of at least 100 mL/kilograms (kg)/year of packed RBC transfusions in the prior 24 months before signing of consent (or the last rescreening for patients going through repeat screening) or, for participants initiating transfusion therapy <24 months before signing of consent, requirement for packed RBC transfusion at least every 3 to 4 weeks for ≥6 months
* Eligible for autologous stem cell transplant as per investigator's judgment.

Key Exclusion Criteria:

* A willing and healthy 10/10 human leukocyte antigen (HLA)-matched related donor is available per investigator's judgement
* Prior hematopoietic stem cell transplant (HSCT)
* Participants with associated α-thalassemia and >1 alpha deletion, or alpha multiplications
* Participants with sickle cell β-thalassemia variant
* Clinically significant and active bacterial, viral, fungal, or parasitic infection as determined by the investigator

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who Achieve Transfusion Independence for at Least 12 Consecutive Months (TI12) | Up to 24 Months After CTX001 Infusion

SECONDARY OUTCOMES:
Proportion of Participants Achieving at Least 95 Percent (%), 90%, 85%, 75% and 50% Reduction in Annualized Transfusions | From Baseline up to 24 Months After CTX001 Infusion
Transfusion Free Duration for Participants who Achieve TI12 | Up to 24 Months After CTX001 Infusion
Proportion of Alleles With Intended Genetic Modification Present in Peripheral Blood Over Time | Up to 24 Months After CTX001 Infusion
Proportion of Alleles With Intended Genetic Modification Present in CD34+ Cells of the Bone Marrow Over Time | Up to 24 Months After CTX001 Infusion
Change in Fetal Hemoglobin Concentration Over Time | From Baseline (Pre-transfusion) up to 24 Months After CTX001 Infusion
Change in Total Hemoglobin Concentration Over Time | From Baseline (Pre-transfusion) up to 24 Months After CTX001 Infusion
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent up to 24 Months After CTX001 Infusion
Proportion of Participants With Engraftment (First day of 3 Consecutive Measurements of Absolute Neutrophil Count [ANC] ≥500 per Microliter [mcgL] on 3 Different Days) | Within 42 Days After CTX001 Infusion
Time to Engraftment | Up to 24 Months After CTX001 Infusion
Incidence of Transplant-related Mortality (TRM) Within 100 Days After CTX001 Infusion | Within 100 Days After CTX001 Infusion
Incidence of TRM Within 12 Months After CTX001 Infusion | Within 12 Months After Infusion
Incidence of All-cause Mortality | From Signing of Informed Consent up to 24 Months After CTX001 Infusion
Relative Reduction in Annualized Volume and Episodes of RBC Transfusions starting Month 10 After CTX001 infusion | From Baseline up to 24 Months After CTX001 Infusion

CONTACTS AND LOCATIONS:
Locations (6):
- TriStar Medical Group Children's Specialists - Pediatric Oncology, Nashville, Tennessee, United States
- Hospital for Sick Children - Hematology, Toronto, Canada
- University Hospital Dusseldorf - Department of Pediatric Oncology, Hematology and Clinical Immunology, Düsseldorf, Germany
- IRCSS Ospedale Pediatrico Bambino Gesu - Dipartimento di Onco-Ematologia e Terapia Cellulare e Genica, Rome, Italy
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - St.Mary's Hospital - Children's Clinical Research Facility, London

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing